CLINICAL TRIAL: NCT05020106
Title: Study on the Diagnostic Cut-off Value of Core Biomarkers in Cerebrospinal Fluid and Blood of Alzheimer's Disease
Brief Title: The Diagnostic Cut-off Value of Core Biomarkers of Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Xiangya Hospital of Central South University (Other); Huashan Hospital (Other); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Jianping Jia, Chief Director, Capital Medical University
Other Study IDs: Biomarker cut-off value
Record Dates: First submitted 2021-07-23; First posted 2021-08-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cerebrospinal fluid,blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Alzheimer's disease: Criteria for AD according to the 2011 NIA-AA
- MCI group: aMCI diagnosed according to the criteria of 2004 Peterson.
- Non-AD dementia: Frontotemporal dementia (FTD); or Parkinson's disease dementia (PDD); or dementia with Lewy bodies (DLB); or vascular dementia (VaD); or corticobasal degeneration (CBD); or dementia not otherwise specified.
- Cognitively normal controls: Individuals with normal cognitive function

SUMMARY:
The participant in this study includes Alzheimer's disease (AD including familial AD and sporadic AD) patients, amnestic mild cognitive impairment (aMCI) patients, non-AD dementia patients and cognitively normal control.

The purpose of this study is to establish the best cut-off value of cerebrospinal fluid (CSF) and blood β-amyloid (Aβ) 42/40, total tau (t-tau) , phosphorylated tau ,inflammatory factors, etc. in diagnosis of Alzheimer's disease (AD).

DETAILED DESCRIPTION:
1. Incorporating patients who meet the criteria from Capital Medical University Xuanwu Hospital including AD, aMCI, non-AD dementia and cognitively normal control.
2. Collect the information of clinical and neuropsychological assessment (mini-mental state examination, MMSE, Montreal cognitive assessment, MoCA, and clinical dementia rating scale, CDR), neuroimaging data including medial temporal atrophy (MTA) score, Fazekas score, MRI, and PET(optional), as well as the biological sample, such as CSF and peripheral blood.
3. To quantify levels of Aβ42, Aβ40, t-tau, p-tau, inflammatory factors, etc. in CSF and blood.
4. Detect all participants ApoE genotype.
5. Independently establish the best cut-off value of Chinese people in our laboratory.
6. Analysis the relationships between core biomarkers in CSF/blood and ApoE genotype and neuroimaging data.
7. Establish combined diagnostic model.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-75. Written informed consent obtained from participant or legal guardian prior to any study-related procedures. The diagnosis of AD is made using the National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria. The diagnosis of aMCI is assigned according to 2004 Petersen criteria. As for non-AD dementia, the McKeith criteria are used for DLB, the revised diagnostic criteria proposed by the International bvFTD Criteria Consortium for behavioral variant FTD, the Gorno-Tempini criteria for the semantic variant FTD or non-fluent aphasia, the Movement Disorder Society Task Force criteria for PDD, the vascular behavioral and cognitive disorders (Vas-Cog) criteria for VaD, the Armstrong's criteria for CBD, the CDC's diagnostic criteria for CJD, etc. In addition, normal cognition is supported by MMSE, CDR and other cognitive function scales.

Exclusion Criteria:

* Other medical or psychiatric illness. No one can serve as an informant. Refused to complete a cognitive test and provide biospecimen.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AD patients (n=800); aMCI patients (n=800);non-AD dementia patients (n=800). cognitively normal controls (n=800);
Sampling Method: Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The cut-off value in diagnosing AD | 1 year
  The best cut-off value of Aβ42, Aβ40, t-tau, p-tau, inflammatory factors, etc. in CSF and blood .
The receiver operating characteristic curve | 1 year
  The receiver operating characteristic curve is used to show the relationship between sensitivity and specificity of core CSF and blood biomarkers in diagnosing AD.
Relationship between biomarker and clinical symptom | 1 year
  The relationship is specifically expressed by relevance

SECONDARY OUTCOMES:
The sensitivity | 1 year
  The sensitivity is used to show the ability of core CSF and blood biomarkers to diagnose AD patients and is represented by true positive/ (true positive +false negative).
The specificity | 1 year
  The specificity is used to show the ability of core CSF and blood biomarkers to avoid false AD patients and rule out AD patients and is represented by true negative/ (false positive + true negative).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jia L, Qiu Q, Zhang H, Chu L, Du Y, Zhang J, Zhou C, Liang F, Shi S, Wang S, Qin W, Wang Q, Li F, Wang Q, Li Y, Shen L, Wei Y, Jia J. Concordance between the assessment of Abeta42, T-tau, and P-T181-tau in peripheral blood neuronal-derived exosomes and cerebrospinal fluid. Alzheimers Dement. 2019 Aug;15(8):1071-1080. doi: 10.1016/j.jalz.2019.05.002. PMID 31422798